CLINICAL TRIAL: NCT07058844
Title: The Effects of a Line Dance Program on Cognitive Function, Physical Function, and Quality of Life in Older Adults With Mild Cognitive Impairment
Acronym: LD-MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wanyu Shu (Other)
Responsible Party: Sponsor-Investigator, Wanyu Shu, Doctor of Philosophy, Hanyang University
Organization: Hanyang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HYU-MCI-2025-01; HYUIRB-202503-002-1 (Other: Hanyang University Institutional Review Board)
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment, Line Dance, Aerobic Exercise, Cognitive Function, BDNF, Dual Task, Older Adults, Quality of Life, Randomized Controlled Trial
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel groups: a high-BPM line dance intervention group, a low-BPM line dance intervention group, or a no-intervention control group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-BPM Line Dance Group (Experimental): Participants in this group will engage in a line dance intervention with music tempos of 130-140 beats per minute (BPM), three times per week for 12 weeks. Each session lasts 60 minutes and includes warm-up, core choreography, and cool-down phases.
  Interventions: Behavioral: High-BPM Line Dance
- Low-BPM Line Dance Group (Experimental): Participants in this group will engage in a line dance intervention with music tempos of 90-100 beats per minute (BPM), three times per week for 12 weeks. Each session lasts 60 minutes and follows the same structure as the HBLD group.
  Interventions: Behavioral: Low-BPM Line Dance
- Control Group (Other): Participants in this group will not receive any specific intervention but will maintain their usual daily activities throughout the 12-week period.
  Interventions: Other: Usual Daily Activity

INTERVENTIONS:
Behavioral: High-BPM Line Dance — A structured aerobic dance program set to music with tempos of 130-140 BPM, designed to improve cognitive and physical function in older adults with MCI.
  Arms: High-BPM Line Dance Group
Behavioral: Low-BPM Line Dance — A structured aerobic dance program set to music with tempos of 90-100 BPM, using the same choreography but slower rhythm and reduced rest intervals.
  Other Names: LBLD
  Arms: Low-BPM Line Dance Group
Other: Usual Daily Activity — No structured intervention will be provided. Participants will continue their routine lifestyle.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the effects of a structured line dance program on cognitive function, physical performance, and quality of life in older women with mild cognitive impairment (MCI). A total of 75 participants aged 60-75 with a diagnosis of MCI will be randomly assigned to one of three groups: a high-beat-per-minute (HBLD) line dance group, a low-beat-per-minute (LBLD) line dance group, or a control group receiving no intervention. The intervention will last for 12 weeks, with sessions held three times per week for 60 minutes. Outcome measures include the Montreal Cognitive Assessment (MoCA), serum brain-derived neurotrophic factor (BDNF), physical function tests, and a quality of life questionnaire. The purpose of this study is to explore the effectiveness of non-pharmacological, rhythm-based exercise interventions for improving cognitive and physical health in older adults with cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged between 60 and 75 years who have been clinically diagnosed with mild cognitive impairment (MCI) at a medical institution (MoCA score ≤ 25)
2. No history of psychiatric disorders
3. Not currently taking any psychiatric medications
4. Normal vision and hearing, and able to complete the assessments without difficulty
5. Physically capable of participating in line dance sessions
6. Provided written informed consent and voluntarily agreed to participate in the study

Exclusion Criteria:

1. Currently taking antidepressants, antipsychotics, or sedative-hypnotic medications
2. Pregnant or potentially breastfeeding
3. Currently participating in another drug-related clinical trial
4. Diagnosed with dementia

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females aged 60 to 75 years are eligible to participate.
Enrollment: 75 (Actual)
Dates: Start 2025-01-19 (Actual); Primary Completion 2025-04-19 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
MoCA | Baseline and 12 weeks post-intervention
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), a validated screening tool for detecting mild cognitive impairment. Scores range from 0 to 30, with higher scores indicating better cognitive performance.
SMS（Sensorimotor Synchronization） | Baseline and after 12-week intervention
  This study used ELAN software (version 6.9) to analyze temporal asynchrony between participants' dance movements and rhythmic cues across four 8-beat sequences (32 beats total). Movement and rhythm layers were time-annotated to assess synchronization accuracy and stability. Data were exported to Excel for analysis. Mean asynchrony indicated synchronization accuracy (higher values = poorer accuracy), while standard deviation reflected synchronization stability (higher values = greater variability)
BDNF (Brain-Derived Neurotrophic Factor) | Baseline and after 12-week intervention
  Serum levels of Brain-Derived Neurotrophic Factor (BDNF) will be measured to assess neuroplasticity-related changes induced by the intervention. Blood samples will be collected, processed, and analyzed using enzyme-linked immunosorbent assay (ELISA). Higher BDNF concentrations are associated with improved synaptic function and cognitive performance.
TUG-cog(Timed Up and Go-Cognitive) | Baseline and after 12-week intervention
  The TUG-cog test will be used to assess dual-task mobility and executive function. Participants are asked to complete the standard Timed Up and Go task while simultaneously performing a cognitive task, such as serial subtraction. The time taken to complete the task is recorded. Longer completion times reflect greater dual-task interference and reduced cognitive-motor integration.
Senior Fitness Test | Baseline and 12 weeks post-intervention
  The Senior Fitness Test (SFT) evaluates physical fitness in older adults across six domains: lower-body strength (30-second chair stand), upper-body strength (30-second arm curl), lower-body flexibility (chair sit-and-reach), upper-body flexibility (back scratch), agility and dynamic balance (8-foot up-and-go), and aerobic endurance (2-minute step test). Higher performance indicates better functional fitness and physical independence.
Short Physical Performance Battery | Baseline and 12 weeks post-intervention
  The Short Physical Performance Battery (SPPB) is a standardized assessment tool used to evaluate lower-extremity physical function in older adults. It consists of three components: balance tests (side-by-side, semi-tandem, and tandem stance), a 4-meter walk test to assess gait speed, and five repeated chair stands to evaluate lower-body strength. The total score ranges from 0 to 12, with higher scores indicating better physical performance and mobility.
Grip Strength | Baseline and 12 weeks post-intervention
  Grip strength will be measured using a digital hand dynamometer (Model EH101, ANTA, Guangdong, China). Participants will stand upright with their arms naturally extended at an angle of approximately 15°-30° from the trunk and will squeeze the device with maximum force for a few seconds. Each hand will be tested twice, and the highest value from either hand will be used for analysis.
Short Form-36 Health Survey | Baseline and 12 weeks post-intervention
  The SF-36 Health Survey is a widely used instrument for evaluating health-related quality of life. It consists of 36 items assessing eight domains: physical functioning, role limitations due to physical and emotional problems, bodily pain, general health, vitality, social functioning, and mental health. Higher scores indicate better perceived health status.

SECONDARY OUTCOMES:
Depression | Baseline and 12 weeks post-intervention
  Depressive symptoms will be assessed using the Geriatric Depression Scale (GDS-15), a validated screening tool for older adults. The scale consists of 15 yes/no questions, with higher scores indicating more severe depressive symptoms.
Blood glucose | Baseline and 12 weeks post-intervention
  asting blood glucose levels will be measured using standard venous blood sampling procedures. The values will be expressed in milligrams per deciliter (mg/dL). Elevated blood glucose levels may indicate impaired glucose metabolism or risk of diabetes.
Berg Balance Scale (BBS) | Baseline and after 12-week intervention
  The Berg Balance Scale (BBS) is a 14-item performance-based measure that assesses static and dynamic balance abilities in older adults. Each item is scored on a 5-point scale ranging from 0 to 4, with a maximum total score of 56. Higher scores indicate better balance ability and lower risk of falling. The BBS is widely used in clinical and research settings to evaluate postural control and balance improvements following intervention.
Blood pressure | Baseline and after 12-week intervention
  Blood pressure will be measured using a calibrated electronic sphygmomanometer. Systolic and diastolic blood pressure will be recorded in a seated position after at least 5 minutes of rest. Measurements will be taken twice, and the average will be used for analysis. Blood pressure is an important indicator of cardiovascular health and may be affected by exercise interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Nankang District Hospital of Traditional Chinese Medicine, Ganzhou, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the participant data and the absence of a secured public data-sharing infrastructure, the individual participant data will not be shared.